CLINICAL TRIAL: NCT02626754
Title: A Prospective Study on Sunitinib as First Line Therapy for Advanced/Metastatic Renal Cell Carcinoma in Asian Population
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: In most sites had difficult to recruitting subjects.
Sponsor: vghtpe user (Other Government)
Responsible Party: Sponsor-Investigator, vghtpe user, Chief, Division of General Urology, Department of Urology, Taipei Veterans General Hospital, Taiwan
Organization: Taipei Veterans General Hospital, Taiwan (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-10-002A
Record Dates: First submitted 2015-12-01; First posted 2015-12-10 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Renal Cell Carcinoma
Keywords: Sunitinib, 2/1 schedule, Renal cell carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sunitinib (Experimental): Sunitinib malate, 12.5mg/capsule, 50mg/day
  Interventions: Drug: Sunitinib malate

INTERVENTIONS:
Drug: Sunitinib malate — Sunitinib 50mg will be given for 2 consecutive weeks then followed by one week of rest.
  Other Names: Sutent

SUMMARY:
This is a multi-national, phase II, single arm study to explore the safety/efficacy and potential biomarkers on sunitinib 2/1 schedule for Asian patients with advanced renal cell carcinoma.

DETAILED DESCRIPTION:
Sunitinib 50mg daily on 4/2 dose schedule has been established as standard of care (SOC) for advanced renal cell carcinoma (RCC). However, Asian patients in real world experienced grade III/IV adverse events much more than expected. This multi-national, phase II, single arm study is going to explore more on the safety/efficacy and relevant biomarkers on sunitinib 2/1 dose schedule in Asian people with advanced RCC.

ELIGIBILITY:
Inclusion Criteria:

* Advanced renal cell carcinoma with histology confirmation
* Grade III/IV AEs happen during first cycle of sunitinib 50mg/day 4 weeks on followed by 2 weeks of rest
* ECOG performance status 0 or 1
* Appropriate vital organ functions

Exclusion Criteria:

* Prior systemic treatment of mRCC
* Patients treated with any neoadjuvant or adjuvant systemic therapy
* Major surgery <4 weeks or radiation therapy <2 weeks of starting the study treatment. Prior palliative radiotherapy to metastatic lesion(s) is permitted, provided there is at least one measurable lesion that has not been irradiated
* Pregnant
* Allergic history to sunitinib

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-08-12 (Actual); Primary Completion 2018-01-02 (Actual); Study Completion 2018-01-02 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (safety and tolerability) | 24 months
  To evaluate the safety and tolerance of sunitinib two weeks on, one week off for advanced renal cell carcinoma

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 24 months
  to evaluate the best response rate of sunitinib 2/1 schedule
progression free survival (PFS) | 24 months
  to evaluate the progression-free survival of sunitinib 2/1 schedule
patient reported outcome (PRO) | 24 months
  to evaluate the change of quality of life with sunitinib 2/1 schedule

OTHER OUTCOMES:
single nuclear polymorphism | 24 months
  to explore the relationship between select SNP associated with sunitinib 2/1 schedule

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Hwa Chang, M.D. Ph.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (7):
- Taiwan (7):
  - Kaohsiung Medical University Chung-HO Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Vterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan

IPD SHARING:
Plan to Share IPD: No